CLINICAL TRIAL: NCT04969952
Title: National Taiwan University Hospital,Taiwan (R.O.C)
Brief Title: Evaluation of an Interventional Module to Assist Physicians Introducing ACP to Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201912238RINA
Record Dates: First submitted 2021-06-29; First posted 2021-07-21 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cancer Patients
Keywords: ACP brochure; Interventional Module; Advance directive; cancer patients

STUDY DESIGN:
Intervention Model Description: Shared decision making (SDM) process through Advance Care Planning (ACP) consultation with cancer patients
Who Masked: Participant, Care Provider
Masking Description: Only investigator know
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A had watching educational module plus ACP brochure
  Interventions: Other: For interventional module
- Group B (Active Comparator): Group B ACP brochure only
  Interventions: Other: For interventional module

INTERVENTIONS:
Other: For interventional module — Using vedio to assist physicians introducing advance care planning to cancer patients

SUMMARY:
Evaluation of an Interventional module to assist physicians introducing ACP to cancer patients

DETAILED DESCRIPTION:
Investigators hypothesize that compared to ACP brochure alone, educational module plus ACP brochure is effective in assisting the physicians to introduce ACP to the patients and completion of AD documentation

ELIGIBILITY:
"Inclusion Criteria" and "Exclusion Criteria"

Inclusion Criteria

1. Older than 20-years-old
2. Diagnosed with cancer
3. Have not signed any form of AD or DNR

Exclusion Criteria

1. Under 20-years-old
2. Can not speak or listen, difficult communication
3. Signed AD or DNR

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Sign DNR (Do-Not-Resuscitate) | 3 month
  After intervention cancer patients willing sing DNR

SECONDARY OUTCOMES:
Completion AD(Advance directive) documentation | 3 month
  After intervention cancer patients completion of a new AD documentation

OTHER OUTCOMES:
Explain and predict health behaviors(Sign DNR / Completion AD) | 3 month
  To evaluate factors that might hinder patient willingness to sign DNR / complete AD documentation by applying the The Transtheoretical Model (TTM).

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yi Cheng Shao-Yi, PHD, Principal Investigator — Shao-Yi Cheng
Locations (2):
- Taiwan (2):
  - Nation Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei County